CLINICAL TRIAL: NCT03414957
Title: Prevalence of Metabolic Syndrome Amongst Malay Women With PCOS
Brief Title: Malay Women With PCOS and Their Association With Metabolic Syndrome
Acronym: MPMSS
Status: Completed | Type: Observational
Sponsor: Cyberjaya University College of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: CRG/05/04/2011; CUCMS/RA/CGS/9-5 (Other Grant/Funding Number: Centre for Graduate Studies, CUCMS)
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Polycystic Ovary Syndrome (PCOS); Metabolic Syndrome
Keywords: Malay women, PCOS, Metabolic Syndrome, Rotterdam criteria
MeSH Terms: conditions — Polycystic Ovary Syndrome; Metabolic Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Serum used for biochemical and genetic tests
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Malay PCOS women: Malay women underwent clinical assessment, followed by pelvic ultrasound scan, biochemical and hormonal blood tests. Using the Rotterdam criteria for the diagnosis of PCOS, Malay women who fulfilled these criteria were inducted into this group. These women were then identified whether they had Metabolic Syndrome or not based on the WHO criteria
  Interventions: Diagnostic Test: Hormonal and biochemical blood tests and ultrasound scanning
- Malay women without PCOS: Malay women underwent clinical assessment, followed by pelvic ultrasound scan, biochemical and hormonal blood tests. Using the Rotterdam criteria for the diagnosis of PCOS, Malay women who did not fulfill these criteria were inducted into this group. These women were then identified whether they had Metabolic Syndrome or not based on the WHO criteria.
  Interventions: Diagnostic Test: Hormonal and biochemical blood tests and ultrasound scanning

INTERVENTIONS:
Diagnostic Test: Hormonal and biochemical blood tests and ultrasound scanning — Subjects undergo clinical assessment, blood tests and a pelvic ultrasound scan, to determine if they have either PCOS or Metabolic Syndrome or both

SUMMARY:
The abnormalities that characterize the Metabolic Syndrome (MetS) confer an increased risk of cardiovascular and other diseases. Women with Polycystic Ovary Syndrome (PCOS), the commonest endocrine disease among women of childbearing age, have an increased risk of developing MetS.

2) The prevalence of MetS in PCOS patients varies among different ethnic groups. Malaysia is a unique country with a multiethnic population. The 3 largest ethnic groups are the Malays, Chinese and Indians. Previous studies in India and China have been able to determine the incidence of PCOS amongst those ethnic groups, but as yet, there is no published data on the prevalence of this disorder amongst women of Malay ethnicity. In this study, I intend to discover the prevalence of MetS amongst Malay women with established PCOS.

DETAILED DESCRIPTION:
Metabolic syndrome (MetS) is a well-known collection of interrelated metabolic conditions that identify patients at increased risk of developing cardiovascular disease. These conditions include diabetes mellitus (DM), high blood pressure, obesity and dyslipidaemia.1 Though the exact pathogenesis of MetS still remains elusive, central obesity and insulin resistance are generally acknowledged as important causative factors. The most recent

International Diabetes Federation (IDF) consensus has developed a definition emphasizing the importance of central obesity with modifications according to ethnic groups.2 Polycystic Ovarian Syndrome (PCOS) is the commonest endocrine disorder in women of reproductive age.3 Around 6-7% of women in the reproductive age group are estimated afflicted with this disorder, which accounts for more than 75% of anovulatory infertility.4 PCOS is characterized by both reproductive and metabolic dysfunctions such as hyperandrogenism, infertility, and increased long term risks of type 2 diabetes, dyslipidaemia, hypertension, visceral obesity, and endometrial cancer. Women with PCOS have been noted to have high incidences of age group-specific prevalence of type 2 DM, myocardial infarct and angina (Mani H 2012). The criteria developed in Rotterdam in 2003 remains the most widely accepted for the diagnosis of PCOS.7 For a diagnosis of PCOS to be made, a minimum of 2 features from oligo/anovulation, hyperandrogenaemia and ultrasound demonstration of polycystic ovaries need to be present. Other causes of polycystic ovaries such as adrenal hyperplasia, androgen-secreting tumours and Cushing's syndrome have to be excluded, of course.

Insulin resistance, which is an established feature of PCOS, leads to compensatory hyperinsulinaemia and affects both the theca and granulosa of the ovary (Franks S 1999, Franks S 2008). Insulin increases serum androgen levels through its function as an ovarian growth hormone (leading to increased theca cell androgen synthesis) and its action on adrenal steroidogenesis (Barbieri RL 1986, Moghetti P 1996). The consequent hyperandrogenaemia interferes with normal folliculogenesis and ovulation. The concerted effects of the elevated serum insulin and androgen levels account for many of the features of PCOS and the metabolic syndrome (Barber TM 2012). It is apparent that insulin resistance, androgen excess, anovulation, metabolic abnormalities and PCOS are all related to each other and form a tangled web. PCOS is now viewed as a clinical phenotype of MetS.5,6

.

ELIGIBILITY:
Inclusion Criteria:

* Malay women aged 20-40 years of age
* clinically healthy and euthyroid (clinically and biochemically) and not on any medication.

Exclusion Criteria:

* women on any hormonal medications

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Malay women
Study Population: Malay women aged 20-40 years of age recruited from the clinical practices of the authors.
  1. These will be subjects attending the Outpatient and the Gynaecology Clinics.
  2. The subjects attending the Gynaecology Clinic will be those presenting with problems achieving pregnancy, excess body hair and/or menstrual disorders.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of Metabolic Syndrome Amongst Malay Women with PCOS | 6 months
  To determine the prevalence of MetS amongst Malay women with PCOS and to compare this prevalence to that amongst Malay women without Polycystic Ovarian Syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Hanif Khan, Principal Investigator — Associate Professor

IPD SHARING:
Plan to Share IPD: Yes
All participant demographics and results as well as calculations
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Once all the data and processing has been completed and will be available until further notice
Access Criteria: Online open